CLINICAL TRIAL: NCT02184819
Title: Effects of Levosimendan Pretreatment in Patients With Low Ejection Fraction (40 % or Less) Undergoing CABG: a Randomised, Double Blind, Multicenter Trial
Brief Title: Preoperative Levosimendan in CABG Patients With Poor LV Function
Acronym: LICORN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P110138
Record Dates: First submitted 2013-10-23; First posted 2014-07-09 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Bypass Grafting; Left Ventricular Dysfonction
Keywords: coronary artery bypass graft; left ventricular dysfunction; low cardiac output syndrome; levosimendan; mortality; inotropic agents; cardiac mechanical assist devices; renal replacement therapy; mechanical ventilation duration; ICU stay
MeSH Terms: conditions — Ventricular Dysfunction, Left; Cardiac Output, Low | interventions — Simendan; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levosimendan (Active Comparator): study drug
  Interventions: Drug: levosimendan
- placebo (Placebo Comparator): placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levosimendan — 24 hour continuous infusion at the rate of 0,1 µg/kg/min
  Other Names: Simdax
  Arms: levosimendan
Drug: Placebo — 24 hour infusion at a rate of 0,1 µg/kg/min assuming that it contains study drug
  Other Names: riboflavine
  Arms: placebo

SUMMARY:
The investigators want to test the hypothesis that an infusion of levosimendan started prior to CABG surgery can reduce incidence and severity of low cardiac output syndrome in patients with poor LV function (EF 40% or less).

DETAILED DESCRIPTION:
Background: Patients with an ejection fraction of less than 40% are at high risk of developing postoperative low cardiac output syndrome (LCOS). Despite the use of potent inotropic agents or even ventricular mechanical assist devices, the mortality rate of such patients remains very high (from 17 to 38%). Their hospital stay is also prolonged and the cost of care for this population is increased. Two studies have suggested that post-operative administration of levosimendan could reduce hospital length of stay and long term (Day180) mortality in patients with LCOS. In addition a few studies have also suggested that pre-operative infusion of levosimendan (pre-conditioning) could reduce the use of other inotropes and mechanical assist devices in patients at high risk of developing LCOS. Unfortunately, the data supporting the beneficial effects of levosimendan in high risk cardiac surgery patients is very limited. Main goal: To evaluate the efficacy of a pre-operative infusion of levosimendan in high risk patients (EF less than 40%) undergoing cardiac surgery (CABG or combined surgery: CABG and valve replacement) to improve outcome. Secondary goals: To evaluate: 1) the clinical safety of a pre-operative infusion of levosimendan, 2) the costs of care in the levosimendan and control groups. Experimental setup: Prospective, multicenter, randomized versus placebo, double-blind trial. Treatment modalities: levosimendan will be administered by the intravenous route, according to a continuous infusion of 0.1mcg/kg/min over 24 hours. Levosimendan infusion (0.1mcg/kg/min) will be started immediately after induction of anaesthesia. The delay between infusion start and skin incision can be estimated between 30 to 60 min. The investigators decided to skip the bolus infusion that is frequently associated with systemic hypotension, which may result in serious adverse events and protocol exclusion. Study duration and patient follow-up: Patients will be recruited over 23 months. Individual follow-up will last 6 months. Overall duration of study will be 29 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* scheduled for CABG with CPB
* with or without asociated cardiac repair
* ejection fraction less than 40%
* signed informed consent

Exclusion Criteria:

* preoperative renal failure (creatinine clearance less than 30 ml/min)
* liver failure (prothrombine time less than 50% in the absence of vitamin K antagonist)
* cardiac surgery without CABG
* pregnancy
* emergency surgery
* known allergy to levosimendan
* severe hypotension prior to surgery
* severe tachycardia
* prior history of torsade de pointe
* dynamic obstruction od left ventricular outflow tract
* lack of signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Confirmed low cardiac output syndrome | within the 28 days after ICU admission
  Composite of the three following items:the need for inotropic agents beyond 24 hours following the end of levosimendan/placebo infusion; the need for post-operative mechanical assist devices (intra-aortic balloon pump: IABP, extra-corporeal life support: ECLS) or failure to wean from these techniques if they were inserted pre-operatively; the need for renal replacement therapy during ICU stay

SECONDARY OUTCOMES:
mortality at Day 28 and Day 180 | 180 postoperative days
The need for inotropic agents beyond 24 hours following the end of levosimendan/placebo infusion | 1 time during 24h beyond operative
The description of renal replacement therapy during ICU stay | within the 28 days after ICU admission
  renal failure requiring renal replacement therapy may occur anytime within 12 hours following surgery and may last 1-2 weeks on average.
number of ventilator-free days and out-of-ICU days at Day 28. | 28 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cholley, MD, PhD, Principal Investigator — Anesthesiology and Intensive Care, Hopital Européen Georges Pompidou, Paris, France; Thibaut Caruba, PharmD, Principal Investigator — Pharmacy department, Hopital Européen Georges Pompidou, Paris, France
Locations (1):
- Hôpital Européen Georges Pompidou, Assistance Publique Hôpitaux de Paris, France, Paris, France

REFERENCES:
- [Background] Levin R, Degrange M, Del Mazo C, Tanus E, Porcile R. Preoperative levosimendan decreases mortality and the development of low cardiac output in high-risk patients with severe left ventricular dysfunction undergoing coronary artery bypass grafting with cardiopulmonary bypass. Exp Clin Cardiol. 2012 Sep;17(3):125-30. PMID 23620700
- [Background] De Hert SG, Lorsomradee S, Cromheecke S, Van der Linden PJ. The effects of levosimendan in cardiac surgery patients with poor left ventricular function. Anesth Analg. 2007 Apr;104(4):766-73. doi: 10.1213/01.ane.0000256863.92050.d3. PMID 17377079
- [Background] Tritapepe L, De Santis V, Vitale D, Santulli M, Morelli A, Nofroni I, Puddu PE, Singer M, Pietropaoli P. Preconditioning effects of levosimendan in coronary artery bypass grafting--a pilot study. Br J Anaesth. 2006 Jun;96(6):694-700. doi: 10.1093/bja/ael082. Epub 2006 Apr 4. PMID 16595616
- [Derived] Cholley B, Caruba T, Grosjean S, Amour J, Ouattara A, Villacorta J, Miguet B, Guinet P, Levy F, Squara P, Ait Hamou N, Carillion A, Boyer J, Boughenou MF, Rosier S, Robin E, Radutoiu M, Durand M, Guidon C, Desebbe O, Charles-Nelson A, Menasche P, Rozec B, Girard C, Fellahi JL, Pirracchio R, Chatellier G; -. Effect of Levosimendan on Low Cardiac Output Syndrome in Patients With Low Ejection Fraction Undergoing Coronary Artery Bypass Grafting With Cardiopulmonary Bypass: The LICORN Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):548-556. doi: 10.1001/jama.2017.9973. PMID 28787507
- [Derived] Caruba T, Hourton D, Sabatier B, Rousseau D, Tibi A, Hoffart-Jourdain C, Souag A, Freitas N, Yjjou M, Almeida C, Gomes N, Aucouturier P, Djadi-Prat J, Menasche P, Chatellier G, Cholley B. Rationale and design of the multicenter randomized trial investigating the effects of levosimendan pretreatment in patients with low ejection fraction (</=40 %) undergoing CABG with cardiopulmonary bypass (LICORN study). J Cardiothorac Surg. 2016 Aug 5;11(1):127. doi: 10.1186/s13019-016-0530-z. PMID 27496105